CLINICAL TRIAL: NCT03910660
Title: Phase 1b/2 Study of BXCL701, a Small Molecule Inhibitor of Dipeptidyl Peptidases, Administered in Combination With the Anti-Programmed Cell Death 1 Monoclonal Antibody Pembrolizumab in Patients With mCRPC Either Small Cell Neuroendocrine Prostate Cancer or Adenocarcinoma Phenotype
Brief Title: A Trial of BXCL701 and Pembrolizumab in Patients With mCRPC Either Small Cell Neuroendocrine Prostate Cancer or Adenocarcinoma Phenotype.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioXcel Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BXCL701-201
Record Dates: First submitted 2019-01-04; First posted 2019-04-10 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Prostate Cancer; Neuroendocrine Tumors; Small Cell Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms; Neuroendocrine Tumors; Carcinoma, Small Cell | interventions — PT-100 dipeptide; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1b (Other): Patients will be observed for dose-limiting toxicity (DLT) during Cycle 1. 3 patients will be treated initially with 0.4 mg BXCL701 plus PEMBRO:
  If there are no DLTs, the dose of BXCL701 will be escalated to 0.6 mg in the next cohort.
  If ≥1/3 of patients has a DLT in Cycle 1, either 3 patients (if 1 experience a DLT) or 6 to 9 patients (if 2 or 3 experiences a DLT) will be added at the 0.4 mg dose.
  At the 0.4mg dose:
  If <1/3 of the patients experience a DLT, consideration will be given to dose to 0.6 mg BXCL701 plus PEMBRO.
  If 1/3 of the patients experience a DLT, the Phase 2a can commence. If >1/3 of the patients experience a DLT, a discussion will be held as to how to proceed.
  Following 0.6 mg dose. If there are no DLTs, the Phase 2a can commence. If ≥1/3 patients have a DLT in Cycle 1, after a discussion, 6 to 9 patients will be added at the 0.6 mg dose.
  For this cohort of 6 to 9 patients:
  If </=1/3 of the patients experience a DLT, the Phase 2a can commence
  Interventions: Drug: BXCL701 plus Pembrolizumab
- Phase 2a (Other): After assessment of the safety and confirmation of the BXCL701/+PEMBRO dose schedule to be used in the subsequent stage, the Phase 2a will begin. Eligible patients will receive BXCL701 QD on Days 1 to 14 of a 21-day cycle plus PEMBRO 200 mg administered IV on Day 1 every 21 days.
  Interventions: Drug: BXCL701 plus Pembrolizumab
- Phase 2b combination (Other): Upon completion of the Phase 2a and achievement of the protocol required composite responses for a given histologic subtype, the Phase 2b enrollment will begin for that subtype. Eligible patients will be randomized to receive:
  • Combination therapy of BXCL701 on Days 1 to 14 of a 21-day cycle plus PEMBRO 200 mg administered IV on Day 1 of every 21 days.
  Interventions: Drug: BXCL701 plus Pembrolizumab
- Phase 2b monotherapy (Other): Upon completion of the Phase 2a and achievement of the protocol required composite responses for a given histologic subtype, the Phase 2b enrollment will begin for that subtype. Eligible patients will be randomized to receive:
  * Monotherapy BXCL701 on Days 1 to 14 of a 21-day cycle. Upon radiographic disease progression with monotherapy, crossover to combination treatment is allowed.
  Interventions: Drug: BXCL701 monotherapy

INTERVENTIONS:
Drug: BXCL701 plus Pembrolizumab — BXCL701 tablets dosage strengths include 0.05mg and 1mg tablets for oral administration.
  BXCL701 will be administered orally as 0.05mg and 1mg tablets. Patients will take the prescribed number of tablets on Days 1 to 14 of each cycle, for a total daily dose of 0.4 mg, 0.6 mg, or an intermediate dose. BXCL701 will be continued until PD or unacceptable toxicity, or closure of the study by the sponsor; no maximum duration of therapy has been set.
  BXCL701 should not be taken on an empty stomach.
  On days when PD studies are being performed, BXCL701 should be administered at the study center and should be administered at approx. the same time of day on each treatment day in the cycle. In cycles in which PD are not evaluated, BXCL701 also should be administered at approx. the same time of day on each treatment day.
  The PEMBRO dose will be 200 mg, administered as an IV infusion over 30 mins. on Day 1 of each 21-day cycle.
  Other Names: BXCL701 plus Pembro
  Arms: Phase 1b; Phase 2a; Phase 2b combination
Drug: BXCL701 monotherapy — BXCL701 tablets dosage strengths include 0.05mg and 1mg tablets for oral administration.
  BXCL701 will be administered orally as 0.05mg and 1mg tablets. Patients will take the prescribed number of tablets on Days 1 to 14 of each cycle, for a total daily dose of 0.4 mg, 0.6 mg, or an intermediate dose. BXCL701 will be continued until PD or unacceptable toxicity, or closure of the study by the sponsor; no maximum duration of therapy has been set.
  BXCL701 should not be taken on an empty stomach.
  On days when PD studies are being performed, BXCL701 should be administered at the study center and should be administered at approx. the same time of day on each treatment day in the cycle. In cycles in which PD are not evaluated, BXCL701 also should be administered at approx. the same time of day on each treatment day.
  Other Names: BXCL701
  Arms: Phase 2b monotherapy

SUMMARY:
An open-label, multicenter, Phase 1b/2 study to identify the recommended Phase 2 dose and assess the efficacy and safety of BXCL701 administered orally, as monotherapy and in combination with PEMBRO, in patients with mCRPC. Patients enrolled in the Phase 2a portion of the study will have either Small Cell Neuroendocrine Prostate Cancer(SCNC)(Cohort A) or adenocarcinoma phenotype (Cohort B), while the Phase 2b randomized portion of the study will enroll only the histologic subtype(s) showing preliminary evidence in Phase 2a. The study will also assess other efficacy parameters, such as rPFS, PSA PFS, OS, and DOR, as well as the safety of the combined treatment. The study will consist of three components.

DETAILED DESCRIPTION:
An open-label, multicenter, Phase 1b/2 study to identify the recommended Phase 2 dose and assess the efficacy and safety of BXCL701 administered orally, as monotherapy and in combination with PEMBRO, in patients with mCRPC. Patients enrolled in the Phase 2a portion of the study will have either Small Cell Neuroendocrine Prostate Cancer(SCNC)(Cohort A) or adenocarcinoma phenotype (Cohort B), while the Phase 2b randomized portion of the study will enroll only the histologic subtype(s) showing preliminary evidence in Phase 2a. The study will also assess other efficacy parameters, such as rPFS, PSA PFS, OS, and DOR, as well as the safety of the combined treatment. The study will consist of three components.

1. Phase 1b: Safety and tolerability of the combination of BXCL701 administered once daily (QD) on Days 1 to 14 of a 21-day cycle plus PEMBRO 200 mg administered intravenously (IV) on Day 1 of every 21 days will be assessed and confirmed in patients with mCRPC. In the first cohort enrolled in the study, the initial dose level of BXCL701 will be 0.4 mg; if there are no safety concerns, this will be escalated to a total daily dose of 0.6 mg.
2. Phase 2a (Simon 2 Stage): Patients will be treated with BXCL701 in combination with PEMBRO. Patients will be grouped in 1 of 2 cohorts based on phenotype.

   * Cohort A: Patients with any Small Cell/Neuroendocrine features, either de novo or treatment-emergent included mixed SCNC.
   * Cohort B: Cohort B: Patients with adenocarcinoma and no evidence of small cell or neuroendocrine features.

Phase 2b (for the histologic subtype[s] showing preliminary efficacy in Phase 2a): Patients within a given subtype will be randomized 2:1 to receive either BXCL701 combined with PEMBRO or BXCL701 monotherapy.

Phase 1b:

Patients will be observed for dose-limiting toxicity (DLT) during Cycle 1. Three patients will be treated initially with BXCL701 0.4 mg plus PEMBRO:

* If there are no DLTs in Cycle 1, the dose of BXCL701 will be escalated to a total daily dose of 0.6 mg in the next cohort of 3 patients.
* If ≥1 of the 3 original patients has a DLT in Cycle 1, after a discussion between the sponsor and the investigator, either 3 patients (if 1 patient experiences a DLT) or 6 to 9 patients (if 2 or 3 patients experiences a DLT) will be added at the 0.4 mg BXCL701 dose level. For this expanded 0.4 mg cohort:

  * If none of the patients experience a DLT, consideration will be given to dose escalation to BXCL701 0.6 mg plus PEMBRO
  * If 1/3 of the patients experience a DLT, the Phase 2 can commence
  * If >1/3 of the patients experience a DLT, a discussion will be held between the investigators and sponsors as to how to proceed.

Following dose escalation to BXCL701 0.6 mg plus PEMBRO in 3 patients:

* If there are no DLTs at this dose level, the Phase 2a can commence.
* If ≥1/3 patients have a DLT in Cycle 1, after a discussion between the sponsor and the investigator, 6 to 9 patients will be added at the 0.6 mg BXCL701 total daily dose level; and consideration of an alternate dosing (e.g., split dose) schedule may be given.
* For this additional cohort of 6 to 9 patients:

  * If </= 1/3 of the patients experience a DLT, the Phase2a can commence.
  * If >1/3 of the patients experience a DLT, consideration will be given to the use of a 0.4 mg total daily dose of BXCL701, or an intermediate dose, plus PEMBRO in the Phase 2a.

ELIGIBILITY:
Inclusion Criteria:

All patients must satisfy the following inclusion and exclusion criteria to be eligible for entry into the trial.

1. Patient has evidence of progressive, metastatic castration-resistant disease, as defined by PCWG3 criteria.

   a. Patients with de novo small cell prostate cancer are not required to have received androgen deprivation therapy (ADT).
2. Progression during or following completion of at least 1 prior line of systemic therapy for locally advanced or metastatic prostate cancer.
3. Phases 2a and 2b Only:

   SCNC - Cohort A of Phase 2a only:
   1. Patient has histologic evidence of SCNC either with archival tissue or a fresh tumor biopsy obtained during screening. Tumor biopsy tissue must be submitted for a central laboratory pathology review; however, enrollment can proceed if SCNC is determined by a local pathology review.
   2. Patient has previously received at least 1 prior line of cytotoxic chemotherapy. Patients who either have refused chemotherapy or are considered unsuitable for chemotherapy may be eligible following discussion with the sponsor.
   3. Must be willing to undergo metastatic tumor biopsy during Screening. Requirement may be waived in patients without safely accessible lesion or for patients with evaluable archival metastatic tumor tissue
   4. Has measurable disease per RECIST 1.1 criteria.

   Adenocarcinoma - Cohort B of Phase 2a; randomized population for Phase 2b
   1. Patient has histologically or cytologically confirmed adenocarcinoma of the prostate without small cell neuroendocrine features.
   2. Patients with soft tissue disease must provide a fresh core or excisional biopsy or archival tissue from a site not previously irradiated for central pathology review; however enrollment may proceed if predominant adenocarcinoma without small cell neuroendocrine features is determined by local pathology review.
   3. Has been treated with at least 1 but no more than 2 second generation AR pathway target agents (e.g., abiraterone acetate and/or enzalutamide or other next generation agent) and at least 1 regimen/line of taxane containing chemotherapy in the mCSPC or mCRPC setting. Patients with known actionable mutations should have progressed on applicable standard care targeted therapy or have documented intolerance to or be unsuitable for such therapy.
   4. RECIST 1.1 measurable disease or detectable bone metastases by whole body bone scintigraphy.
4. Patient has serum testosterone <50 ng/dL during Screening except for those with de novo small cell prostate cancer.

   a. Patients with treatment-emergent SCNC without a history of bilateral orchiectomy are required to remain on luteinizing hormone-releasing hormone (LHRH) analog during the course of protocol therapy except for patients with de novo small cell prostate cancer.
5. Patient has Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
6. Patient is ≥18 years of age.
7. Patient's acute toxic effects of previous anticancer therapy have resolved to ≤Grade 1 except for Grade 2-3 peripheral neuropathy or any grade of alopecia.
8. Patient has adequate baseline organ function, as demonstrated by the following:

   1. Serum creatinine ≤1.5 times institutional upper limit of normal (ULN) or calculated creatinine clearance >50 mL/min;
   2. Serum albumin ≥2.5 g/dL;
   3. Total bilirubin ≤1.5 × ULN;
   4. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 × institutional ULN (patients with hepatic metastases must have AST/ALT ≤5 × ULN).
9. Patient has adequate baseline hematologic function, as demonstrated by the following:

   1. Absolute neutrophil count (ANC) ≥1.5 × 109/L.
   2. Hemoglobin ≥8 g/dL and no red blood cell transfusions during the prior 14 days.
   3. Platelet count ≥100 × 109/L and no platelet transfusions during the prior 14 days.
10. Male patients and their female partners of childbearing potential must agree and commit to use a barrier contraception throughout the duration of the study until at least 6 months following the last dose of study drug, in addition to their female partners using either an intrauterine device or hormonal contraception and continuing until at least 6 months following the last dose of study drug. This criterion may be waived for male patients who have had a vasectomy >6 months before signing the informed consent form.

    Exception: In the United States, female partners of study participants are not required to use contraception as a condition of their partners' eligibility, but female partners with child bearing potential should consider use of effect methods of contraception for the duration of their male partners' study participation and for at least 6 months following the last dose of study medication.
11. Patient has signed informed consent prior to initiation of any study-specific procedures or treatment.
12. Patient is able to adhere to the study visit schedule and other protocol requirements, including follow-up for overall survival (OS).

Exclusion Criteria:

1. Patient has received treatment with >2 cytotoxic chemotherapy regimens for castration-resistant prostate cancer (CRPC). Chemotherapy in the hormone-sensitive setting does not count in this assessment provided the last dose was >6 months before study entry. A change in chemotherapy agents due to intolerance after brief exposure may not count in this assessment, pending review with Medical Monitor.
2. Patient has received external-beam radiation or another systemic anticancer therapy within 14 days or 5 half-lives, whichever is shorter, prior to study treatment.
3. Patient has received treatment with an investigational systemic anticancer agent within 14 days prior to study drug administration.
4. Patient has received prior treatment with an anti-PD-1, anti-PD-L1, anti-programmed death ligand 2 (PD-L2) agent or with an agent directed to another co-inhibitory T-cell receptor (e.g., cytotoxic T lymphocyte-associated antigen 4 [CTLA-4], OX-40, CD137) or requires concomitant treatment with DPP4 inhibitors.
5. Patient has an additional active malignancy that may confound the assessment of the study endpoints. If the patient has a past cancer history (active malignancy within 2 years prior to study entry) with substantial potential for recurrence, this must be discussed with the sponsor before study entry. Patients with the following concomitant neoplastic diagnoses are eligible: non-melanoma skin cancer and carcinomas in situ (including transitional cell carcinoma, anal carcinoma, and melanoma in situ).
6. Patient has clinically significant cardiovascular disease (e.g., uncontrolled or any New York Heart Association Class 3 or 4 congestive heart failure, uncontrolled angina, history of myocardial infarction, unstable angina or stroke within 6 months prior to study entry, uncontrolled hypertension or clinically significant arrhythmias not controlled by medication).
7. QT interval corrected for heart rate using Bazett's formula (QTcB) >480 msec at Screening.
8. Patient has uncontrolled, clinically significant pulmonary disease (e.g., chronic obstructive pulmonary disease, pulmonary hypertension) that in the opinion of the investigator would put the patient at significant risk for pulmonary complications during the study.
9. Patient has brain or leptomeningeal metastases that are symptomatic and progressive on imaging. Patients with a history of central nervous system (CNS) metastases must have received appropriate treatment. Central nervous system imaging is not required prior to study entry unless there is a history of CNS involvement or clinical suspicion of CNS involvement. Imaging of patients with a prior history of CNS metastases should be compared to prior imaging to discern disease progression.
10. Patient has an active autoimmune disease or Grade ≥3 non-infectious pneumonitis that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) or treatment with drugs (e.g., neomercazol, carbimazole) that function to decrease the generation of thyroid hormone by a hyperfunctioning thyroid gland (e.g., in Graves' disease) is not considered a form of systemic treatment of an autoimmune disease.
11. Patient has a diagnosis of immunodeficiency or is receiving systemic steroid therapy at a prednisone equivalent dose of >10 mg daily for at least 1 week or other form of immunosuppressive therapy within 7 days prior to Cycle 1 Day 1 (C1D1).
12. Patient has uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, suspected or active SARS-CoV-2 (COVID-19) infection, disseminated intravascular coagulation, or psychiatric illness/social situations that would limit compliance with study requirements.
13. Patient has known positive status for human immunodeficiency virus, active or chronic Hepatitis B, or Hepatitis C. Screening is not required.
14. Patient has any medical condition which, in the opinion of the investigator, places the patient at an unacceptably high risk for toxicity.
15. Any dysphagia, odynophagia, esophageal dysmotility or stricture, known GI malabsorption syndrome, or intractable diarrhea that may significantly alter the absorption of orally administered study drug.
16. Patients with history of symptomatic orthostatic hypotension within 3 months prior to enrollment. Orthostatic hypotension is defined as a drop in systolic blood pressure (BP) of ≥ 20 mmHg or diastolic BP of ≥ 10 mmHg with assumption of an upright posture.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2024-12-12 (Actual)

PRIMARY OUTCOMES:
Phase 2a: Estimate the composite response rate of the combination of BXCL701 + PEMBRO | up to 36 months
  Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 criteria; circulating tumor cell (CTC) conversion from >5/7.5 mL to <5/7.5 mL per Veridex assay; and 50% or greater prostate-specific antigen (PSA) decline from baseline.
Phase 2b: Evaluate response rates in patients treated with the combination of BXCL701 + PEMBRO and with BXCL701 monotherapy | up to 36 months
  To evaluate the response rates, defined by RECIST 1.1 criteria, by histologic subtype in patients treated with the combination of BXCL701 + PEMBRO and with BXCL701 monotherapy.

SECONDARY OUTCOMES:
Phase 2a: Estimate the median radiographic progression-free survival (rPFS) of the combination of BXCL701 and PEMBRO in Cohort A and B | up to 36 months
  The median time frame with progression-free survival with the use of BXCL701 in combination with Pembro determined by radiographic evidence.
Phase 2a: Estimate the median PSA progression-free survival (PSA PFS) of the combination of BXCL701 and PEMBRO in Cohort A and B. | up to 36 months
  The median time frame with progression-free survival with the use of BXCL701 in combination with Pembro
Phase 2a: Estimate the median overall survival (OS) of the combination of BXCL701 and PEMBRO in Cohort A and B. | up to 36 months
  The median time frame with overall survival with the use of BXCL701 in combination with Pembro
Phase 2a: Estimate the median duration of response (DOR) of the combination of BXCL701 and PEMBRO in Cohort A and B. | up to 36 months
  The timeframe in which the tumor reacts to BXCL701 in combination with Pembro
Phase 2a: Determine the risk profile of the use of BXCL701 in combination with PEMBRO. | up to 36 months
  Determines the frequency and severity of known and unknown adverse events with the use of BXCL701 in combination with Pembro
Phase 2a: Assess population pK of BXCL701 | Up to 36 months
  To assess the population pharmacokinetics of BXCL701 using sparse pharmacokinetic sampling.
Phase 2a: Assess pharmacodynamic profile of BXCL701 and Pembro | Up to 36 months
  To assess the pharmacodynamic profile of the combination of BXCL701 and PEMBRO by measuring relevant effects on those cytokines previously shown to be modulated by BXCL701 in humans.
Phase 2b: Estimate the CRR, OS, duration response, rPFS and PSA PFS of the BXCL701+Pembro. | Up to 36 months
  To estimate the CRR, OS, duration of response, rPFS, and PSA PFS of the BXCL701 + PEMBRO combination and monotherapy in Cohort A and B, respectively. Composite response rate is defined as achieving 1 or more of the following:
  * Objective response by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria
  * 50% or greater PSA decline from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Amir Hafeez, MD, Study Director — Bioxcel Therapeutics; Vincent O'Neill, MD, Study Chair — Bioxcel Therapeutics
Locations (12):
- United States (9):
  - University of California San Francisco (UCSF), San Francisco, California
  - BioXcel Clinical Research Site, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - Moffitt Cancer Center and Research Institute, Tampa, Florida
  - BioXcel Clinical Research Site, Detroit, Michigan
  - Center for Advanced Medicine / R.J. Zuckerberg Cancer Center (Northwell Health Cancer Institute), Lake Success, New York
  - Weill Cornell Medicine New York, New York, New York
  - White Plains Hospital Center for Cancer Care, White Plains, New York
  - The Ohio State University, Columbus, Ohio
- United Kingdom (3):
  - BioXcel Clinical Research Site, Glasgow, England
  - BioXcel Clinical Research Site, London, Great Britain
  - BioXcel Clinical Research Site, Sutton, Surrey

IPD SHARING:
Plan to Share IPD: No